CLINICAL TRIAL: NCT02472821
Title: Test of Hearing Health Education Programs for Farm and Rural Youth
Acronym: FARMYOUTHEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Progressive Agriculture Foundation (Unknown)
Responsible Party: Principal Investigator, Marjorie McCullagh, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F037851-00; R01DC013885 (NIH)
Record Dates: First submitted 2015-06-09; First posted 2015-06-16 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Noise-induced Hearing Loss
MeSH Terms: conditions — Hearing Loss, Noise-Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Interactive Lesson (Active Comparator): Subjects will receive a community-based face-to-face interactive youth educational program on hearing health
  Interventions: Behavioral: Interactive youth educational program
- Interactive lesson + Web-based booster (Active Comparator): Subjects will receive a community-based face-to-face interactive youth educational program on hearing health followed by an Internet-based educational booster
  Interventions: Behavioral: Interactive youth educational program; Behavioral: Internet-based educational booster
- No-intervention control (No Intervention): No interventions; pre- and post- measures only.

INTERVENTIONS:
Behavioral: Interactive youth educational program — Participation in a community-based face-to-face interactive youth educational program focusing on hearing health (i.e., noise hazards, risk of noise-induced hearing loss, mechanism of injury to the internal ear, and preventive measures)
  Other Names: Progressive Agriculture Foundation Safety Days
  Arms: Interactive Lesson; Interactive lesson + Web-based booster
Behavioral: Internet-based educational booster — Visit to an educational Web site focused on hearing health
  Other Names: Dangerous Decibels Virtual Exhibit
  Arms: Interactive lesson + Web-based booster

SUMMARY:
Farm and rural youth have frequent exposure to hazardous noise on the farm and recreationally, and have an increased prevalence of noise-induced hearing loss (NIHL). There is a lack of programs to prepare this high-risk population to use hearing conservation strategies. This randomly-controlled trial of innovative community-based interventions is designed to compare effectiveness and sustainability of approaches to increase youths' use of hearing conservation strategies. Consistent use of hearing conservation strategies is expected to reduce rates of NIHL and other negative effects of high noise exposure, and improve quality of life in this high-risk and underserved group.

DETAILED DESCRIPTION:
Farm and rural youth have frequent exposure to hazardous noise on the farm and recreationally, and have an increased prevalence of noise-induced hearing loss. An estimated 2 million children and adolescents younger than 20 years of age are exposed to farm noise hazards as farm residents, farm family workers, hired workers, children of migrant or seasonal workers, or farm visitors. This noise exposure begins from an early age, and is compounded by frequent exposure to recreational noise (e.g., all-terrain vehicles and firearms). Farm youth also have an increased prevalence of noise-induced hearing loss, a permanent and irreversible condition negatively impacting quality of life of the affected person, as well as their family members.

Although primary prevention offers the best opportunity for success, farm and rural youth are rarely served by an Occupational Safety and Health Administration-mandated or other hearing conservation program. Although previous tests of limited educational programs to promote hearing conservation among small groups of farm youth have demonstrated short-term increases in hearing protector use (or intent to use), their impact on this population has been limited by program reach and sustainability.

The purpose of this project is to test innovative hearing health education programs delivered to a large target group and to determine the effectiveness and sustainability of these programs in promoting hearing health among farm and rural youth. Specifically, this project includes: a) an interactive Safety Days program alone, b) an interactive Safety Days program followed by an Internet-based booster, and c) a no-intervention control. This test is designed to determine the most effective and sustainable approach to hearing health education among farm and rural youth. Only with effective and sustainable hearing health education programs can use of hearing conservation strategies be increased to prevent noise-induced hearing loss and other negative effects of high noise exposure, and improve quality of life in this high-risk and under-served group.

This project will involve a partnership between the University of Michigan School of Nursing and a major farm and rural youth safety education organization to accomplish project aims.

This randomized-controlled trial of innovative community- based interventions is designed to determine the most effective and sustainable approach to increase youths' use of hearing protection strategies. Results of this study will be used to inform future research-to-practice studies to protect the health and safety of farm and rural youth. Consistent use of hearing conservation strategies is expected to reduce rates of noise-induced hearing loss and other negative effects of high noise exposure, and improve quality of life in this high-risk and underserved group.

ELIGIBILITY:
Inclusion Criteria:

* enrollment in grade 4
* parental consent
* English speaking
* attending a Safety Days event included in the cluster sampling

Exclusion Criteria:

* (none)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2093 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
Self-reported use of hearing conservation strategies (i.e., using hearing protection devices, walking away from hazardous noise, or turning down sources of hazardous noise) when in high noise | 12 months

SECONDARY OUTCOMES:
Cost effectiveness | 12 months
  Costs association with program delivery (i.e., instruction time, travel time)
Sustainability | 12 months
  Key stakeholders' ratings of program capacity to maintain program and its benefits over time using scale prepared for this purpose

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie C McCullagh, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] McCullagh MC, Banerjee T, Yang J. Protocol of a test of hearing health education programs for farm and rural youth. BMC Public Health. 2015 Oct 16;15:1061. doi: 10.1186/s12889-015-2393-y. PMID 26475373